CLINICAL TRIAL: NCT04418440
Title: Nutritional Treatment for the Amelioration of Traumatic Brain Injury
Acronym: NUTRA-TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 273132
Record Dates: First submitted 2020-05-14; First posted 2020-06-05 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Routine NHS care following traumatic brain injury
- Treatment (Experimental): Routine NHS care following traumatic brain injury plus daily dose of test compound (oral nutritional supplement)
  Interventions: Dietary Supplement: Souvenaid oral nutritional supplement (Nutricia)

INTERVENTIONS:
Dietary Supplement: Souvenaid oral nutritional supplement (Nutricia) — Daily dose of a commercially available oral nutritional supplement based around the active compound recipe Fortasyn Connect, produced by Nutricia, Danone.
  Arms: Treatment

SUMMARY:
To test the feasibility of administering a commercially available neurotrophic oral nutritional supplement (ONS) for adult patients with acute traumatic brain injury at the Royal London Hospital.

DETAILED DESCRIPTION:
The study will be a randomised controlled non-blinded trial of adult patients with acute traumatic brain injury at the Royal London Hospital.

There will be randomisation to one of two non-blinded trial groups:

1. Usual standard NHS care (control group)
2. Usual standard NHS care plus daily oral dose of Souvenaid® ONS

The trial protocol will commence between 3-7 days after admission. The trial timeline provides a summary of intervention and assessments.

The trial will last 12 months. The first 6 months will be the formal trial with two groups and follow up assessments. This will be performed on intention to treat basis. After this initial phase the investigators will provide an opportunity for all participants from either group (control or treatment) to take Souvenaid® ONS for a further 6 months with a clinical follow up appointment.

ELIGIBILITY:
Inclusion Criteria:

* Adult between 18 yrs and 80 yrs of age
* Acute traumatic brain injury with confirmed radiological features

Exclusion Criteria:

* Allergies to fish oil/milk/soya
* Medical history of galactosaemia
* Non-traumatic aetiology to head injury
* Unable to receive enteral nutrition
* Craniectomy during admission (loss of integrity of skull convexity)
* Concurrent active neurological disease
* Pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility to conduct the protocol as stated | 10 months
  To assess logistical issues which might prevent a fully powered study being carried out using this protocol. The investigators will primarily be looking at retention rate. If there is an attrition rate of over 80% then this protocol will be deemed not feasible.

SECONDARY OUTCOMES:
Brain network connectivity | 10 months
  As measured by resting state EEG
Cognitive function | 10 months
  Changes to cognitive function as measure by CANTAB-TBI cognitive test. This is a validated and widely used clinical tool for cognitive assessment in TBI and assesses cognition using the following battery of tests (range of scores in brackets with lower score being worse performance and higher being better performance): paired associates learning (0-70); reaction time (100-5100); spatial working memory (0-153); multitasking test (0-160); one touch stockings of Cambridge (0-15).
Plasma phospholipid levels | 10 months
  Plasma phospholipid levels will be measured using thin layer chromatography and/or LC-MS. Batch analysis
Omega-3 index | 10 months
  The omega-3 index will be analysed in red blood cells. Therefore, lipids will be extracted from red blood cells, followed by transesterification and quantification using gas chromatography coupled to a flame ionisation detector.
Neurofilament light levels | 10 months
  Plasma or serum neurofilament light levels will be measured using either a commercially available enzyme-linked immunosorbent assay, a commercially available chemi-luminescent assay, or the commercially available SIMOA assay. Combined samples will be run on each plate to account for inter plate variability.
Inflammatory markers | 10 months
  Inflammatory markers such as cytokines will be analysed using either enzyme-linked immunosorbent assays or a multiplex system. Combined samples will be run on each plate to account for inter plate variability.
C-reactive protein | 10 months
  CRP will be measured independently using an enzyme-linked immunosorbent assay. Combined samples will be run on each plate to account for inter plate variability

CONTACTS AND LOCATIONS:
Overall Officials: Chris Uff, Principal Investigator — Barts Health
Locations (1):
- Bart Health, Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not applicable, not part of protocol